CLINICAL TRIAL: NCT03578224
Title: Contrast-Enhanced Ultrasound Identification of Sentinel Nodes in Esophageal Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F.235; R21CA218946 (NIH); JT 12449 (Other: JeffTrial Number)
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Esophagus
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Biopsy, Fine-Needle; Sonazoid; perfluorobutane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (EUS, FNA, perflubutane microbubble) (Experimental): Participants undergo standard of care unenhanced endoscopic ultrasound (EUS) and fine needle aspiration (FNA) of identified lymph nodes. Participants then receive perflubutane microbubble peri- or intratumorally and undergo contrast-enhanced EUS followed by FNA of identified lymph nodes.
  Interventions: Procedure: Endoscopic Ultrasound-Guided Fine-Needle Aspiration (EUS-FNA); Procedure: Contrast-Enhanced Ultrasound; Procedure: Fine-Needle Aspiration; Drug: Sonazoid (Perflubutane)

INTERVENTIONS:
Procedure: Endoscopic Ultrasound-Guided Fine-Needle Aspiration (EUS-FNA) — Undergo EUS-FNA
Procedure: Contrast-Enhanced Ultrasound — Undergo CEUS
Procedure: Fine-Needle Aspiration — Undergo FNA
Drug: Sonazoid (Perflubutane) — Sonazoid (ultrasound contrast agent) will be injected in 0.25 mL increments at 12, 3, 6, and 9 o'clock positions around the tumor using a 19 - 22 gauge needle system under EUS guidance

SUMMARY:
This pilot trial studies how well an ultrasound with a contrast agent (perflubutane microbubble [Sonazoid]) works in identifying sentinel lymph nodes in participants with esophageal cancer. Sentinel lymph nodes are lymph nodes to which the cancer is likely to spread from the primary tumor. Diagnostic procedures, such as contrast-enhanced ultrasound, may work better in identifying sentinel lymph nodes and finding out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the accuracy of contrast-enhanced endoscopic lymphosonography guided fine-needle aspiration (FNA) of sentinel lymph nodes compared with unenhanced endoscopic ultrasonography (EUS) guided FNA in the characterization of esophageal cancer-associated lymph nodes using pathology as the reference standard.

SECONDARY OBJECTIVES:

I. To assess the ability of contrast-enhanced endoscopic lymphosonography guided FNA compared with unenhanced EUS guided FNA in the overall detection of biopsy proven cancer-involved sentinel lymph nodes.

II. To assess the impact of overall tumor staging by contrast-enhanced endoscopic lymphosonography compared with unenhanced EUS.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with esophageal cancer.
* Be scheduled for staging endoscopic ultrasound with the intent for lymph node evaluation.
* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.
* Be medically stable.
* If a female and pre-menopausal, must have a negative pregnancy test.

Exclusion Criteria:

* Females who are pregnant or nursing.
* Patients with other primary cancers requiring systemic treatment.
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable.
* Patients with known hypersensitivity or allergy to any component of Sonazoid.
* Patients with cardiac shunts or unstable cardiopulmonary conditions.
* Patients with congenital heart defects.
* Patients with severe emphysema, pulmonary vasculitis, pulmonary hypertension, respiratory distress syndrome, or a history of pulmonary embolism.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Accuracy rate of traditional endoscopic ultrasonography (EUS) with suspicious node biopsy and lymphosonography for sentinel node identification | Up to 2 years
  The number and locations of the nodes identified by the two imaging approaches (contrast-enhanced ultrasound [CEUS] and unenhanced EUS) will be compared using McNemar's test for correlated proportions as well as using a one-sided t-test with a Wilcoxon non-parametric adjustment (normal distribution will be tested) with pathology as the reference standard for sentinel lymph node detection and considering exact binomial p-values less than 0.05 to be significant. The findings of lymphosonography will be correlated to pathological findings (including degree of metastatic involvement) to determine sensitivity and specificity and the rate of cancerous nodes identified by CEUS relative to those of unenhanced EUS using a clustered conditional logistic regression analysis of correlated proportions (equivalent to a clustered McNemar's test).

SECONDARY OUTCOMES:
Number of nodes identified | Up to 2 years
  The number and locations of the nodes identified by the two imaging approaches (CEUS and unenhanced EUS) will be compared using McNemar's test for correlated proportions as well as using a one-sided t-test with a Wilcoxon non-parametric adjustment (normal distribution will be tested) with pathology as the reference standard for sentinel lymph node detection and considering exact binomial p-values less than 0.05 to be significant. The findings of lymphosonography will be correlated to pathological findings (including degree of metastatic involvement) to determine sensitivity and specificity and the rate of cancerous nodes identified by CEUS relative to those of unenhanced EUS using a clustered conditional logistic regression analysis of correlated proportions (equivalent to a clustered McNemar's test).

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Bin Liu, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/